CLINICAL TRIAL: NCT05164276
Title: Effect of Head Position on Nasotracheal Intubation With Video-laryngoscope in Pediatric Patients: A Randomized Controlled Trial
Brief Title: Head Position on Pediatric Nasotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, yun jeong chae, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AJIRB-MED-INT-21-432
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Intubation
MeSH Terms: interventions — Head-Down Tilt

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sniffing group (Active Comparator): Before intubation, the patient's shoulder is supported by a 5cm pillow to make neck flexion with extension of atlanto-occipital joint, confirming that the external auditory meatus and sternal notch plane are horizontal and aligned. Then, nasotracheal intubation is performed with a reinforced tube (Mallinckrodt Medical, Dublin, Ireland) using video-laryngoscope (AceScope, AceMedical, Seoul, Korea).
  Interventions: Other: Head position
- Neutral group (Experimental): Before intubation, the patient's head is placed without a pillow on the bed. Then, nasotracheal intubation is performed with a reinforced tube (Mallinckrodt Medical, Dublin, Ireland) using video-laryngoscope (AceScope, AceMedical, Seoul, Korea).
  Interventions: Other: Head position
- Flexed group (Experimental): Before intubation, the patient's neck is flexed with pads until the chin touches the chest. Then, nasotracheal intubation is performed with a reinforced tube (Mallinckrodt Medical, Dublin, Ireland) using video-laryngoscope (AceScope, AceMedical, Seoul, Korea).
  Interventions: Other: Head position

INTERVENTIONS:
Other: Head position — Before nasotracheal intubation, patient's head is positioned to one of three positions according to assigned group: sniffing, neutral or flexed position.

SUMMARY:
The aim of study is to evaluate whether the head position facilitates pediatric nasotracheal intubation when using a video-laryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-8 years old
* Amerian Society of Anesthesiologists I or II
* Patients who need nasotracheal intubation for surgery

Exclusion Criteria:

* A recent airway infection within 14 days
* Anatomical deformity in head and neck
* Modified Mallampati score IV
* Bleeding tendency in preoperative laboratory examination

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Intubation time | Within 5 minutes
  The time between entry of the nasotracheal tube into a nostril and appearance of a carbon dioxide wave on the monitor.

SECONDARY OUTCOMES:
Intubation difficulty scale | During intubation
  The sum of score from seven variables including intubation attempts, supplementary operators, the use of alternative techniques, glottic exposure, the lifting force applied during laryngoscopy, the necessity of applied external laryngeal pressure, and position of vocal cords.
  From 0 (easiest) to 8 (most difficult)
Epistaxis score | When removing the video-laryngoscope
  grade 1 (no-epistaxis), grade 2 (mild, blood on the tube only), grade 3 (moderate, blood pooling in the pharynx), or grade 4 (severe: blood impedes intubation)
Numeric rating scale of intubation difficulty | During intubation
  Subjective intubation difficulty from 0 (easiest) to 10 (most difficult)

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University School of Medicine, Suwon, Gyeonggi-do, South Korea